CLINICAL TRIAL: NCT06193317
Title: Effects of taVNS on Fibromyalgia Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Felipe Fregni, MD, PhD, MPH, Director of Spaulding Neuromodulation Center, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023P003467
Record Dates: First submitted 2023-12-21; First posted 2024-01-05 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Fibromyalgia, Pain
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active taVNS (Experimental): TaVNS will be administered by an earset, with conductive eartips placed on the auricular concha of the ears, connected to a stimulator, and during active stimulation, we stimulate both the cymba conchae and external auditory canal of both left and right ears with the following parameters: 30Hertz (Hz), 200-250 us, and with adjustable intensity for 60 min for 16 sessions.
  Interventions: Device: Transauricular vagus nerve stimulation (taVNS)
- Sham taVNS (Sham Comparator): Sham condition will have the same device, with an earset, and conductive eartips placed in the same location of the active stimulation; however during 60 min for 16 sessions there will be no current and the device will be turned off.
  Interventions: Device: Transauricular vagus nerve stimulation (taVNS)

INTERVENTIONS:
Device: Transauricular vagus nerve stimulation (taVNS) — Transauricular vagus nerve stimulation (taVNS) is a simple technique in which small surface electrodes are placed over the skin of the ear that are thought to be innervated by the auricular branch of the vagus nerve (ABVN).

SUMMARY:
Transauricular vagus nerve stimulation (taVNS) is a newer delivery system, using a non-invasive stimulation device placed at the ear's concha. TaVNS is a portable, safe, and low-cost intervention, and according to some studies, taVNS may influence nociception and pain perception, which can lead to potential applications for various painful illnesses, including fibromyalgia (FM). This trial aims to investigate the clinical effects of taVNS on pain control in FM subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Older than 18 years old.
2. Diagnosis of FM pain according to the American College of Rheumatology (ACR) 2010 criteria (existing pain for more than six months with an average of at least 3 on a 0-10 VAS scale).
3. must have the ability to feel sensation by Von-Frey fiber on the forearm.
4. Able to provide informed consent to participate in the study.

Exclusion Criteria:

1. Subjects who have unstable medical conditions (e.g., uncontrolled diabetes, uncompensated cardiac issues, heart failure, or chronic obstructive pulmonary disease) or who have functional deficits, as self-reported.
2. history of substance abuse within the past six months as self-reported (if the subject reports a history of substance abuse, we will confirm using the Diagnostic and Statistical Manual of Mental Disorders (DSM-V) criteria).
3. Presence of implanted cranial electronic medical devices (e.g., cochlear implants).
4. pregnancy (as the safety of taVNS in the pregnant population (and children) has not been assessed (though the risk is non-significant), we will exclude pregnant women (and children). Women of child-bearing potential will be required to take a urine pregnancy test during the screening process and every two weeks of stimulation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2028-05-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
pain severity using the Brief Pain Inventory (BPI pain) | From Baseline to Visit 19 (at 4 weeks)
  Brief Pain Inventory (BPI) is a short self-assessment questionnaire that provides information on various dimensions of pain including how pain developed, the types of pain a patient experiences, time of day pain is experienced, as well as current ways of alleviating pain. The BPI also includes the Visual Analog Scale (VAS) Pain scale, a simple 10-point scale (0 = ''no pain'', 10 = ''pain as bad as you can imagine'') measuring patients' pain, on average and at the present time. The BPI provides information on pain intensity (the sensory dimension) and the degree to which pain interferes with function (the reactive dimension).

CONTACTS AND LOCATIONS:
Locations (1):
- Spaulding Hospital Cambridge, Cambridge, Massachusetts, United States

REFERENCES:
- [Result] Kim AY, Marduy A, de Melo PS, Gianlorenco AC, Kim CK, Choi H, Song JJ, Fregni F. Safety of transcutaneous auricular vagus nerve stimulation (taVNS): a systematic review and meta-analysis. Sci Rep. 2022 Dec 21;12(1):22055. doi: 10.1038/s41598-022-25864-1. PMID 36543841
- [Result] Parente J, Carolyna Gianlorenco A, Rebello-Sanchez I, Kim M, Mario Prati J, Kyung Kim C, Choi H, Song JJ, Fregni F. Neural, Anti-Inflammatory, and Clinical Effects of Transauricular Vagus Nerve Stimulation in Major Depressive Disorder: A Systematic Review. Int J Neuropsychopharmacol. 2024 Mar 1;27(3):pyad058. doi: 10.1093/ijnp/pyad058. PMID 37870480
- [Result] Gianlorenco ACL, de Melo PS, Marduy A, Kim AY, Kim CK, Choi H, Song JJ, Fregni F. Electroencephalographic Patterns in taVNS: A Systematic Review. Biomedicines. 2022 Sep 6;10(9):2208. doi: 10.3390/biomedicines10092208. PMID 36140309
- [Result] Molero-Chamizo A, Nitsche MA, Bolz A, Andujar Barroso RT, Alameda Bailen JR, Garcia Palomeque JC, Rivera-Urbina GN. Non-Invasive Transcutaneous Vagus Nerve Stimulation for the Treatment of Fibromyalgia Symptoms: A Study Protocol. Brain Sci. 2022 Jan 12;12(1):95. doi: 10.3390/brainsci12010095. PMID 35053839